CLINICAL TRIAL: NCT04241263
Title: Feasibility Study of a Neonatal Wireless Transmission System (NeWTS)
Brief Title: Neonatal Wireless Monitoring System for Intensive Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Kathryn Beardsall, University Lecturer, Consultant Neonatologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: A095011
Record Dates: First submitted 2020-01-12; First posted 2020-01-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Preterm Infant; Infant, Newborn; Low; Birthweight, Extremely (999 Grams or Less)
Keywords: Patient monitoring; Medical device; Wireless
MeSH Terms: conditions — Premature Birth; Birth Weight

STUDY DESIGN:
Masking Description: This is a feasibility study but there are two arms and the babies, parents and staff will all be considered participants -it will be approximately 20 families recruited
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparative assessment of data quality (Other): Quantitative comparison between the current wired system and the new wireless system
  Interventions: Device: Wireless vital sign monitoring - comparative
- Usability (Other): Qualitative assessment of the new wireless system
  Interventions: Device: Wireless vital sign monitoring - usability

INTERVENTIONS:
Device: Wireless vital sign monitoring - comparative — Participants who currently have vital sign monitoring will, in addition, have the wireless system attached. We will then collect up to 24 hours of vital sign data from both systems, which will allow us to make direct comparisons between them.
  Arms: Comparative assessment of data quality
Device: Wireless vital sign monitoring - usability — Babies will be recruited who do not currently require vital sign monitoring. The wireless system will be attached to these babies by nurses who have been trained in its use. A parent will then be asked to perform Kangaroo Care for as long as they feel comfortable. After the baby is placed back in its cot, and the sensors have been removed, we will conduct (separate) interviews with the nurse and the parent on the neonatal intensive care unit (NICU).
  Arms: Usability

SUMMARY:
Babies who require intensive care need to have their heart rate, oxygen levels and temperature measured continuously using specially designed monitors. These monitors allow the clinical team to constantly assess the baby and see if they are becoming unwell. However, these monitors each have separate wires to connect them to the baby. Another important part of care in these babies is being able to allow parents to hold their babies, getting them out of their incubators to be cuddled. This is called Kangaroo care and has been shown to impact on long term health for both babies and parents.

We have designed a system to free babies of the wires that tether them to the monitors. This system has been tested in adults and we now want to test them on the babies.

There are two study parts with two different questions:

1. How good is the data? This will compare the new wireless system with the existing system. Babies will have both standard wired monitors and the new wireless monitor on at the same time so we can compare the data to see how good is the quality of the data collected on the new system.
2. What do parents and staff think about the wireless system during Kangaroo care? Babies who no longer need monitoring (but who previously had been monitored with the wired system), will have the wireless system attached and the parent will take their baby from the cot for Kangaroo Care. After the baby has been placed back in the cot, we will conduct interviews with the parent and the nurse to find out what they thought of the new system.

We hope this will help the investigators to understand about how good the data is we collect and how we might be able to improve the system.

DETAILED DESCRIPTION:
Summary of study design

This is a single-center study recruiting from the neonatal intensive care unit (NICU) at Addenbrooke's Hospital, Cambridge. There are 2 study parts:

1. Quantitative assessment of the accuracy of the new system in comparison with standard clinical monitoring systems
2. Qualitative Assessment of parent and staff views of caring for babies with the new system in comparison with conventional clinical monitoring systems

Quantitative study arm Study population Up to 24 participants will be recruited from the Addenbrooke's Hospital NICU. The participants will be recruited from three groups, defined by the BAPM Categories of Care The population size has been selected to include sufficient babies to collect a reasonable amount of data to ascertain, with confidence, our defined outcomes. Furthermore, the data should come from across the range of variables seen in babies requiring intensive care while limiting exposure of the infants at most risk. The study will be performed in a stepwise fashion, starting with those infants requiring lower dependency care.

Inclusion criteria

* Babies being cared for on the NICU at Addenbrookes Hospital
* Written, informed parental consent Exclusion criteria
* Known to have an intolerance to silicone or silicone gel adhesives.
* Has a pacemaker or other implanted electronic device.

Planned procedures Participants will have the newly developed wireless sensors for ECG, pulse oximetry, and temperature attached adjacent to the current clinical, wired sensors. Once the application sites have been identified and prepared, the sensors will be placed on the baby by an appropriately trained individual. The wireless receiver will connect to a separate patient monitor to log the comparative data. This study monitor will be covered and silenced such that data will not be visible to the clinical team, and it will not be possible to confuse the study monitor from the 'clinical' monitor. The sensors will be in place for a period of up to 24 hours. After this period, the study sensors will be removed, and the site inspected by a member of the research team and scored using the standard tissue viability scoring system already in use on the unit. The sensors will be disposed of in keeping with the unit and Trust policy.

After the study intervention, a questionnaire will be given to the nurse caring for the baby to determine their views on the wireless system.

Data collection Data will be collected from both the study monitor and the 'clinical' monitor. The data are formed of two types: parameter data and waveform data. Parameter data has a two-second interval. The waveform data has a period of approximately 4ms.

Qualitative study arm

Study population Up to 10 participants will be recruited from the Addenbrooke's Hospital. This is in line with other studies with similar cohorts and balances the need to obtain a range of views and experiences, with the imposition on parents' time in such an environment.

Inclusion criteria

* BAPM level transitional care babies who do not clinically require vital sign monitoring.
* The baby has had vital sign monitoring at some point during their stay on the unit.
* Written, informed parental consent Exclusion criteria
* Known to have an intolerance to silicone or silicone gel adhesives.
* Has a pacemaker or other implanted electronic medical device.

Planned procedure Babies who are not indicated for vital sign monitoring will have the wireless monitoring system attached. Once the application sites have been identified and prepared, the sensors will be placed on the baby by an appropriately trained individual. The wireless receiver will connect to the study monitor to log the vital sign data, and all alarms will be silenced. The monitor will be covered and silenced such that it will not impact on clinical care.

The baby will be transferred from the cot/incubator to the parent for kangaroo care as per standard NICU procedure. The parent and baby will remain in contact for as long as the parent is comfortable, and the baby remains stable and in keeping with unit policy and procedures. The baby will then be transferred back to the cot, and monitoring will be removed.

Semi-structured interviews lasting approximately 30 minutes will then be conducted with, (i) the nurse, and (ii) the parent(s). These interviews will focus on previous experiences with vital sign monitoring systems, and their experience of using the new wireless system.

ELIGIBILITY:
Inclusion Criteria:

(i) Babies being cared for on the NICU at Addenbrooke's Hospital (ii) Written, informed parental consent

Exclusion Criteria:

(i) Known to have an intolerance to silicone or silicone gel adhesives. (ii) Has a pacemaker, or other implanted electronic device

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean (SD) difference in ECG waveform data | Up to 24 hours of monitoring data per participant
  comparison of data between wired (standard care) and wireless system

SECONDARY OUTCOMES:
Impact on care: qualitative interviews with parents and staff | immediately post intervention
  Qualitative interviews
Impact on care: qualitative questionnaire with parents and staff | immediately post intervention
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: kathryn beardsall, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No